CLINICAL TRIAL: NCT07361354
Title: A Phase 1, Randomized, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of AGA2118 in Healthy Japanese, Chinese, and Caucasian Participants
Brief Title: A Phase 1 Ethnobridging TriaL of AGA2118 in Healthy Japanese, Chinese, and Caucasian ParticipantS (ATLAS)
Acronym: ATLAS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Angitia Incorporated Limited (Industry)
Responsible Party: Sponsor
Organization: Angitia Biopharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT24-006
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants; Pharmacokinetic Study
Keywords: Ethnobridging; Healthy volunteer

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Japanese) (Experimental): One of three single ascending dose cohorts of healthy Japanese participants. Participants will receive a single administration of low dose AGA2118.
  Interventions: Drug: AGA2118
- Cohort 2 (Japanese) (Experimental): One of three single ascending dose cohorts of healthy Japanese participants. Participants will receive a single administration of medium dose AGA2118.
  Interventions: Drug: AGA2118
- Cohort 3 (Japanese) (Experimental): One of three single ascending dose cohorts of healthy Japanese participants. Participants will receive a single administration of high dose AGA2118.
  Interventions: Drug: AGA2118
- Cohort 4 (Caucasian) (Experimental): Healthy Caucasian participants will receive a single administration of high dose AGA2118.
  Interventions: Drug: AGA2118
- Cohort 5 (Chinese) (Experimental): Healthy Chinese participants will receive a single administration of high dose AGA2118.
  Interventions: Drug: AGA2118

INTERVENTIONS:
Drug: AGA2118 — Participants will receive AGA2118 administered by subcutaneous injection

SUMMARY:
This study will evaluate the effects of a single dose of AGA2118 in Japanese, Chinese, and Caucasian participants

DETAILED DESCRIPTION:
This Phase 1 ethnobridging study will evaluate the pharmacokinetics, pharmacodynamics, and safety of AGA2118 in Japanese, Chinese, and Caucasian participants. Participants will be administered AGA2118 at the start of the study and followed for 85 days. Eighteen Japanese participants will be enrolled and randomized 1:1:1 to one of three doses of AGA2118 to be administered at a single timepoint. Following completion of dosing of the Japanese participants, 6 Caucasian participants will be enrolled to receive the highest dose at a single timepoint. They will be matched to Japanese participants (group average matching) by sex and weight. Additionally, 6 Chinese participants will be enrolled to receive a single administration of the highest dose. These participants may be enrolled at any time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, aged 18 to 65 years
* 25-hydroxyvitamin D ≥30 ng/mL and agree to taking calcium and vitamin D supplements during the study
* Meet the criteria for Japanese, Chinese, or Caucasian ethnicity

Exclusion Criteria:

* Participating or have participated in another clinical trial within the past 6 months
* Any bone fracture within the past 6 months
* History of myocardial infarction or stroke within the past 12 months
* Malignancy within the past 5 years
* Current hyper- or hypocalcemia
* Pregnant or breastfeeding women, or women planning to become pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | Day 1 to up to the end of study (85 days post-dose)
  Cmax of AGA2118 after dosing
Time to maximum concentration (Tmax) | Day 1 to up to the end of study (85 days post-dose)
  Tmax of AGA2118 after dosing
Area under the concentration-time curve (AUC) | Day 1 to up to the end of study (85 days post-dose)
  AUC of AGA2118 after dosing
Half-life (t1/2) | Day 1 to up to the end of study (85 days post-dose)
  t1/2 of AGA2118 after dosing
Clearance (CL) | Day 1 to up to the end of study (85 days post-dose)
  CL of AGA2118 after dosing
Volume of distribution (Vd) | Day 1 to up to the end of study (85 days post-dose)
  Vd of AGA2118 after dosing

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | Baseline to the end of study (85 days post-dose)
  Occurrence of TEAEs

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles EPCU, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No